CLINICAL TRIAL: NCT02741076
Title: A Randomized, Double-blind, Placebo-controlled, Clinical Trial of Structured Opioid Discontinuation Versus Continued Opioid Therapy in Suboptimal and Optimal Responders to High-dose Long-term Opioid Analgesic Therapy for Chronic Pain.
Brief Title: Discontinuation vs Continuation of Long-term Opioid Therapy in Suboptimal and Optimal Responders With Chronic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit sufficient no. of subjects over an acceptable time period
Sponsor: Member Companies of the Opioid PMR Consortium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2065-5
Record Dates: First submitted 2016-02-10; First posted 2016-04-18 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Opioid-Related Disorders; Opiate Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Structured discontinuation opioid therapy Suboptimal Responder (Experimental)
  Interventions: Drug: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER); Drug: Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)
- Structured discontinuation opioid therapy Optimal responders (Experimental)
  Interventions: Drug: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER); Drug: Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)
- Continuation of opioid therapy Suboptimal responders (Experimental)
  Interventions: Drug: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER); Drug: Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)
- Structured Continuation of opioid therapy Optimal responders (Experimental)
  Interventions: Drug: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER); Drug: Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)

INTERVENTIONS:
Drug: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER) — Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)
Drug: Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER) — Continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER)

SUMMARY:
The purpose of this study is to evaluate the effect on pain intensity (PI) of structured discontinuation of long-term opioid analgesic therapy compared to continuation of opioid therapy in Suboptimal and Optimal Responders to high-dose, long-term opioid analgesic therapy for chronic low back pain (CLBP).

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled study which consisted of a common Screening Visit for all subjects, then different schedules for Optimal and Suboptimal Responders, followed by a common schedule for the Blinded Structured Opioid Discontinuation Period (BSODP) and Follow-up Period.

The original protocol (10 Jan 2016) was amended twice: Amendment 1 (07 Jul 2016) and Amendment 2 (08 Feb 2017). Screening of subjects only started after Amendment 1 approval. Approximately half the subjects were screened under Amendment 1 and half under Amendment 2. The original statistical analysis plan (SAP) was amended twice as well based on the protocol amendments. The current SAP is version 1.3, dated 11 April 2018, which added a section to list the analyses that were not being completed as a result of the premature termination of this study.

The duration of the entire study for each subject was approximately 33 to 37 weeks. For Suboptimal Responders: the study duration included Screening Period of up to 3 weeks, Run-in Period of 1 week, Baseline Period of 1 week, Blinded Structured Opioid Discontinuation Period of 24 weeks, and Follow-up Period of 4 weeks.

For Optimal Responders: the study duration included Screening Period of up to 3 weeks, Observation Period of 1 week, Taper Period up to 2 weeks, Open Label Titration Period of 3 weeks, Blinded Structured Opioid Discontinuation Period of 24 weeks, and Follow-up Period of 4 weeks.

The primary endpoint was the change in the mean Average PI score on the 0-10 Numerical Ratings Scale (NRS) from Baseline to the 1 week period before the Week 12 visit. Data were summarized using descriptive statistics (number of observations [n], mean, standard deviation, median, first and third quartiles, minimum, and maximum for continuous variables; and frequency and percentage for categorical variables). Due to the inability to recruit a sufficient number of subjects over an acceptable period of time, the study was terminated prematurely and efficacy analyses were reduced and only a brief summary of the statistical analyses of the primary endpoint in each group (Suboptimal Responders and Optimal Responders) were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or non-pregnant, non-lactating female aged 18 to 75 years, inclusive.
2. Have a clinical diagnosis of non-radicular CLBP (pain that occurs in an area with boundaries between the lowest rib and the crease of the buttocks) of Class 1 or proximal radicular (above the knee) pain of Class 2 based on the Quebec Task Force Classification for Spinal Disorders (subjects with previous surgery or chronic pain syndrome, i.e., classes 9.2 or 10, will be allowed if their pain does not radiate or radiates only proximally) for a minimum of 12 months and

   1. For the Suboptimal Responder group, pain must have been present for at least several hours a day and have an Average PI score of 6-9 on an 11-point NRS within the past 24 hours of screening.
   2. For the Optimal Responder group, subjects must have an Average PI score of 1-4 on an 11-point NRS within the past 24 hours of screening.
3. Have been taking ER/LA opioids or immediate release opioids (at least 4 times at day) for at least 12 months.
4. Have been taking one of the 3 index ER opioid drugs around-the-clock at a twice-a-day frequency for at least 3 consecutive months at a total daily dose within the range shown below.

   Daily Dose Range
   1. Morphine sulfate extended-release: 120-540mg
   2. Oxycodone extended-release: 80-360mg
   3. Oxymorphone extended-release: 40-180mg
5. Be considered, in the opinion of the Investigator, to be in generally good health other than CLBP at screening based upon the results of a medical history, physical examination, 12-lead ECG, and laboratory profile.
6. Speak, read, write, and understand English (to reduce heterogeneity of data), understand the consent form, and be able to effectively communicate with the study staff.
7. Have access to the Internet (to access the patient support program).
8. Voluntarily provide written informed consent.
9. Be willing and able to complete study procedures.

Exclusion Criteria:

1. Have any clinically significant condition that would, in the opinion of the Investigator, preclude study participation or interfere with the assessment of pain and other symptoms of CLBP or increase the risk of opioid-related AEs.
2. Have a primary diagnosis of fibromyalgia, complex regional pain syndrome, neurogenic claudication due to spinal stenosis, spinal cord compression, acute nerve root compression, severe or progressive lower extremity weakness or numbness, bowel or bladder dysfunction as a result of cauda equina compression, diabetic amyotrophy, meningitis, diskitis, back pain because of secondary infection or tumor, or pain caused by a confirmed or suspected neoplasm.
3. Have undergone a surgical procedure for back pain within 6 months prior to the Screening Visit.
4. Have had a nerve or plexus block, including epidural steroid injections or facet blocks, within 1 month prior to the Screening Visit or botulinum toxin injection in the lower back region within 3 months prior to screening.
5. Have a history of confirmed malignancy within past 2 years, with exception of basal cell or squamous cell carcinoma of the skin that has been successfully treated.
6. Have uncontrolled blood pressure, i.e., subject has a sitting systolic blood pressure >180 mm Hg or <90 mm Hg, or a sitting diastolic blood pressure >110 mmHg or <40 mm Hg at screening.
7. Have a body mass index (BMI) >45 kg/m2. Anyone with a BMI >40 but <45 will complete a screening tool (STOPBang Questionnaire) to rule out high risk of obstructive sleep apnea.
8. Have clinically significant depression based on a score of ≥20 on the Patient Health Questionnaire (PHQ-8)
9. Have suicidal ideation associated with actual intent and a method or plan in the past year: "Yes" answers on items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS).
10. Have a previous history of suicidal behaviors in the past 5 years: "Yes" answer (for events that occurred in the past 5 years) to any of the suicidal behavior items of the C-SSRS.
11. Have any lifetime history of serious or recurrent suicidal behavior. (Non-suicidal self-injurious behavior is not a trigger for a risk assessment unless in the Investigator's judgment it is indicated.)
12. Have clinically significant abnormality in clinical chemistry, hematology or urinalysis, including serum glutamic-oxaloacetic transaminase/aspartate aminotransferase or serum glutamic pyruvic transaminase/alanine aminotransferase ≥3 times the upper limit of the reference range or a serum creatinine >2 mg/dL at screening.
13. Have severe enough psychiatric or substance abuse disorder to compromise the subject's safety or scientific integrity of the study.
14. Have on-going litigation associated with back pain or pending applications for workers compensation or disability issues or subjects who plan on filing litigation or claims within the next 12 months; subjects with settled past litigations will be allowed as will subjects who have been on workers compensation or disability claims for at least 3 months.
15. Have used a monoamine oxidase inhibitor within 14 days prior to the start of study medication.
16. Are taking agonist-antagonists (pentazocine, butorphanol or nalbuphine), buprenorphine, methadone, barbiturates, or more than one type of benzodiazepine within 1 month prior to screening.
17. Have a positive urine drug test (UDT) for illicit drugs (including marijuana), non-prescribed controlled substances (opioid or non-opioid), or alcohol at screening.
18. Have taken any investigational drug within 30 days prior to the Screening Visit or are currently enrolled in another investigational drug study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (61):
  - G & L Research, Foley, Alabama
  - Horizon Research Partners, Mobile, Alabama
  - Healthscan Clinical Trials, Montgomery, Alabama
  - Center for Pain and Supportive Care, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Quality of Life Medical and Research Centers, Tucson, Arizona
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Aviva Research, Escondido, California
  - Global Clinical Trials, Irvine, California
  - The Helm Center for Pain Management, Laguna Woods, California
  - Alexander Ford, MD, Los Angeles, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Catalina Research Institute, Montclair, California
  - North Country Clinical Research, Oceanside, California
  - Westview Clinical Research, Placentia, California
  - Foothills Pain Management Clinic, Pomona, California
  - Northern California Research, Sacramento, California
  - Breakthrough Clinical Trials, San Bernardino, California
  - Optimus Medical Group, San Francisco, California
  - Mountain View Clinical Research, Denver, Colorado
  - Care Research Center, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Eastern Research, Hialeah, Florida
  - Finlay Medical Research, Miami, Florida
  - Future Clinical Research, Miami, Florida
  - South Florida Clinical Research, Miami, Florida
  - Empire Clinical Research, Miami Lakes, Florida
  - Martin E Hale, MD, Plantation, Florida
  - Florida Medical Pain Management, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Sestron Clinical Research, Marietta, Georgia
  - Healthcare Research Network II, Blue Island, Illinois
  - Indiana Pain and Spine Clinic, South Bend, Indiana
  - Mid-American Psysiatrists, Overland Park, Kansas
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Oakland Medical Research, Troy, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - St Louis Clinical Trials, St Louis, Missouri
  - Red Rock Clinical Research, Las Vegas, Nevada
  - OnSite Clinical Solutions, Mooresville, North Carolina
  - Clinical Trials of America, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Medical Research International, Oklahoma City, Oklahoma
  - SP Research, Oklahoma City, Oklahoma
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Founders Research Corporation, Philadelphia, Pennsylvania
  - Carolina Center for Advanced Management of Pain, Spartanburg, South Carolina
  - Healthy Concepts, Rapid City, South Dakota
  - Comprehensive Pain Specialists, Hendersonville, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Biopharma Informatic Research Center, Houston, Texas
  - Coastal Medical Group, Houston, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Interventional Pain and Spine Specialists, Chester, Virginia
  - Healing Hands of Virginia, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit 14 September 2016; Date of Early Study Termination 29 January 2018
Pre-assignment Details: Prior to randomization, subjects gave consent and entered a pre-assignment period that assessed eligibility for the intervention phase of the study.
Groups:
- Structured Discontinuation Opioid Therapy Suboptimal Responder: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER) Suboptimal Responder
- Continuation of Opioid Therapy Suboptimal Responder: Structured continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Suboptimal Responder
- Structured Discontinuation Opioid Therapy Optimal Responder: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Optimal Responder
- Continuation of Opioid Therapy Optimal Responder: Structured continuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Optimal Responder
Period: Overall Study
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Started | 13 | 12 | 3 | 4
Completed | 10 | 7 | 1 | 2
Not Completed | 3 | 5 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Sponsor Request | 2 | 3 | 0 | 1
Not completed — No additional information available | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Structured Discontinuation Opioid Therapy Suboptimal Responder: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Suboptimal Responder
- Total: Total of all reporting groups
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder | Total
Number analyzed (Participants) | 13 | 12 | 3 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 3 | 4 | 28
  >=65 years | 1 | 3 | 0 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 56.5 [31 to 75] | 56.1 [35 to 75] | 41.7 [29 to 52] | 49.8 [35 to 58] | 54.1 [29 to 75]
Age, Customized [Count of Participants; unit: Participants]
  <25 | 0 | 0 | 0 | 0 | 0
  25-49 | 3 | 4 | 2 | 1 | 10
  50-64 | 9 | 5 | 1 | 3 | 18
  Equal to or greater than 65 | 1 | 3 | 0 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 1 | 2 | 18
  Male | 5 | 5 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 1 | 2 | 12
  Not Hispanic or Latino | 8 | 8 | 2 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 0 | 1 | 8
  White | 8 | 10 | 3 | 3 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 3 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Average Pain Intensity (PI) Score on the 0-10 Numerical Ratings Scale (NRS)
Description: Baseline is defined as the mean of the available Average PI scores on the 0-10 Numerical Ratings Scale (NRS) over the 7-day Baseline Period. For the scheduled post-randomization visits, mean Average Pain Intensity is defined as the means of the respective PI scores over the 7 days preceding the visit. If there is only one daily PI score available, the mean is not calculated, and the data point is considered missing.
  PI = Pain Intensity. Higher scores indicate more pain intensity; lower scores less pain intensity. Scale range 0-10.
Time Frame: From baseline to the 1 week period prior to the Week 12 visit
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale | -0.2198 (0.83544) | -0.3328 (1.00514) | 0.3750 (1.28794) | 1.00 (0.00)

2. Secondary Outcome: Change in Mean Average Pain Intensity Score (PI) Score on the 0-10 Numerical Ratings Scale (NRS)
Description: as for outcome 1
Time Frame: From baseline to weeks 4, 8, 16, 20, and 24
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale
  4 weeks: number analyzed (Participants) | 12 | 9 | 2 | 4
  4 weeks | -0.1123 (0.77962) | -0.1413 (0.99386) | 0.4940 (0.64818) | 0.3143 (0.38951)
  8 weeks: number analyzed (Participants) | 12 | 9 | 2 | 3
  8 weeks | -0.3671 (0.86810) | 0.0984 (0.62794) | 0.3393 (0.63135) | 0.1413 (0.25046)
  16 weeks: number analyzed (Participants) | 10 | 7 | 2 | 3
  16 weeks | -0.3462 (0.79086) | -0.5714 (1.37382) | -0.6964 (1.38896) | 0.4508 (0.48807)
  20 weeks: number analyzed (Participants) | 9 | 6 | 2 | 2
  20 weeks | -0.4153 (0.81486) | -0.6873 (1.08941) | -0.4821 (1.08591) | -0.3095 (0.03367)
  24 weeks: number analyzed (Participants) | 10 | 6 | 1 | 1
  24 weeks | -0.5000 (0.83692) | -0.1532 (1.23299) | 0.2857 (NA) — Not estimable due to single subject in group | 1.5 (NA) — Not estimable due to single subject in group

3. Secondary Outcome: Number of Suboptimal Responders With Pain Intensity (PI) Score Improvement Relative to Baseline PI Measured on the 0-10 Numerical Ratings Scale (NRS)
Description: Percent pain intensity difference (PID) relative to baseline is defined as 100* ((baseline Average PI - mean Average PI at visit)/baseline Average PI). The percentages are based on number of subjects in the Intent-to-Treat set per treatment group. PI is measured on the Numerical Ratings Scale (NRS). Higher scores indicate more pain intensity; lower scores less pain intensity. Scale range 0-10.
  This outcome measure applies only to Suboptimal Responders.
Time Frame: Weeks 12 and 24
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 0 | 0
Participants
  greater than or equal to 30% Week 12 | 1 | 0 | 0 | 0
  greater than or equal to 20% Week 12 | 1 | 1 | 0 | 0
  greater than or equal to 10% Week 12 | 3 | 3 | 0 | 0
  >0% (any improvement) Week 12 | 7 | 5 | 0 | 0
  greater than or equal to 30% Week 24 | 0 | 0 | 0 | 0
  greater than or equal to 20% Week 24 | 1 | 1 | 0 | 0
  greater than or equal to 10% Week 24 | 5 | 3 | 0 | 0
  >0% (any improvement) Week 24 | 8 | 3 | 0 | 0

4. Secondary Outcome: Number of Suboptimal Responders With Pain Intensity (PI) Score Worsening Relative to Baseline PI Measured on the 0-10 Numerical Ratings Scale (NRS)
Description: Percent pain intensity difference (PID) relative to baseline is defined as 100* ((baseline Average PI - mean Average PI at visit)/baseline Average PI). The percentages are based on number of subjects in the Intent-to-Treat set per treatment group. PI is measured on the Numerical Ratings Scale (NRS). Higher scores indicate more pain intensity; lower scores less pain intensity. Scale range 0-10.
  This outcome measure applies only to Optimal Responders.
Time Frame: Weeks 12 and 24
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Structured Discontinuation Opioid Therapy Optimal Responders: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Optimal Responder
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responders | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 0 | 0 | 3 | 4
Participants
  greater than or equal to 40% Week 12 | 0 | 0 | 1 | 0
  Greater than or equal to 30% Week 12 | 0 | 0 | 1 | 0
  greater than or equal to 20% Week 12 | 0 | 0 | 1 | 2
  Greater than or equal to 10% Week 12 | 0 | 0 | 1 | 2
  Equal to 0% (any worsening) Week 12 | 0 | 0 | 1 | 2
  Greater than or equal to 40% week 24 | 0 | 0 | 0 | 0
  greater than or equal to 30% Week 24 | 0 | 0 | 0 | 1
  greater than or equal to 20% Week 24 | 0 | 0 | 0 | 1
  Greater than or equal to 10% Week 24 | 0 | 0 | 1 | 1
  Greater than 0% (any worsening) Week 24 | 0 | 0 | 1 | 1

5. Secondary Outcome: Change From Baseline on Sleep Quality Measured by Medical Outcomes Study (MOS)
Description: The MOS Sleep Scale is a 12-item questionnaire which measures sleep quality in 7 scales over the past 4 weeks: sleep disturbance, snoring, sleep short of breath or headache, sleep adequacy, sleep somnolence, and 2 sleep problems indexes. In addition, the average hours of sleep over the past 4 weeks is recorded as a raw measure and also coded as an optimal sleep index.
  The MOS is scored and the sleep scales calculated according to the MOS Sleep Scale User's Manual v1.0 (Spritzer and Hays, 2003). The scores on the dimensions and the sleep indices were converted to a 0-100 scale, with higher scores reflecting more of the attribute implied by the name (e.g. greater sleep disturbance, greater sleep adequacy of sleep).
Time Frame: Weeks 12 and 24
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale
  Sleep Disturbance Week 12 | -5.673 (18.5378) | -5.00 (35.3754) | -0.417 (8.3229) | 2.813 (16.5635)
  Snoring Week 12 | 0.00 (37.42) | 10.00 (27.63) | 0.00 (40.00) | 15.00 (19.15)
  Awaken Short of Breath or Headache Week 12 | 3.1 (21.36) | 0.00 (26.97) | 13.3 (23.09) | 10.00 (11.55)
  Sleep Adequacy Week 12 | 10.00 (18.26) | 0.8 (24.29) | 3.3 (25.17) | 5.00 (19.15)
  Sleep Somnolence Week 12 | -4.6154 (20.43683) | 2.7778 (25.33945) | 6.6667 (17.63834) | 8.3333 (14.78237)
  Sleep Problems Index I Week 12 | -4.1026 (12.25907) | -0.2778 (16.66414) | 4.4444 (12.61980) | 0.8333 (9.95360)
  Sleep Problems Index II Week 12 | -5.4274 (13.32784) | -2.222 (15.63651) | 2.0370 (15.23816) | 1.8056 (12.50823)
  Sleep Quantity Week 12 | 0.1 (0.95) | -0.1 (1.31) | -2.3 (2.89) | 0.5 (0.58)
  Sleep Disturbance Week 24 | 5.375 (18.4283) | -10.313 (12.4418) | -5.00 (14.1421) | -10.000 (3.7500)
  Snoring Week 24 | 0.0 (42.16) | 0.0 (38.54) | 40.00 (28.28) | 13.3 (11.55)
  Awaken Short of Breath or Headache Week 24 | 10.0 (34.32) | 10.0 (41.40) | 20.0 (28.28) | 40.00 (40.00)
  Sleep Adequacy Week 24 | 0.0 (35.28) | 13.8 (19.23) | 25.0 (21.21) | 0.00 (20.00)
  Sleep Somnolence Week 24 | 6.0000 (33.47378) | -4.1667 (24.92847) | 16.6667 (32.99832) | -11.1111 (7.69800)
  Sleep Problems Index I Week 24 | 6.6667 (25.09242) | -9.1667 (20.91176) | -6.6667 (18.85618) | -2.2222 (11.70628)
  Sleep Problems Index II Week 24 | 4.8333 (22.91520) | -6.8056 (17.25100) | -2.2222 (21.99888) | -2.2222 (6.40698)
  Sleep Quantity Week 24 | -0.8 (1.81) | -0.1 (1.46) | 0.5 (0.71) | 0.0 (0.00)

6. Secondary Outcome: Participants Sleep Quantity Measured by Medical Outcomes Study (MOS)
Description: Optimal Sleep Index is based on the average number of hours of sleep each night during the past 4 weeks. Index=1 represents 7-8 hours and Index=0 represents < 7 hours or > 8 hours.
Time Frame: 4 weeks prior to baseline and prior to 12 and 24 week visits
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Participants
  Index=0 Baseline | 10 | 9 | 2 | 3
  Index=1 Baseline | 3 | 3 | 1 | 1
  Index=0 Week 12 | 11 | 10 | 2 | 1
  Index=1 Week 12 | 2 | 2 | 1 | 3
  Index=0 Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Index=0 Week 24 | 9 | 7 | 1 | 2
  Index=1 Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Index=1 Week 24 | 1 | 1 | 1 | 1

7. Secondary Outcome: Change From Baseline in the Patient Health Questionnaire Depression Scale (PHQ-8)
Description: The PHQ-8 is an 8-item questionnaire that aims at assessing the level of mood of a subject. Each item is scored from 0 = "not at all" to 3= "nearly every day"; the total score, which is the sum of the score for each item, can be from 0 to 24. A score ≥10 is considered major depression and ≥20 is severe major depression.
Time Frame: Weeks 12 and 24
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale
  12 Weeks | -1.2 (4.75) | -0.8 (4.94) | 3.3 (6.81) | 3.3 (6.50)
  24 Weeks | 0.7 (3.47) | -1.1 (3.98) | 0.00 (7.07) | -1.3 (0.58)

8. Secondary Outcome: Number of Participants Reporting Major or Severe Major Depression Using Patient Health Questionnaire Depression Scale (PHQ-8)
Description: The PHQ-8 is an 8-item questionnaire that aims at assessing the level of depression of a subject. Each item is scored from 0 = "not at all" to 3= "nearly every day"; the total score, which is the sum of the scores for each item, can be from 0 to 24. A score >= 10 is considered major depression and >= 20 is severe major depression.
Time Frame: Baseline, 12 and 24 week visit
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Participants
  Major Depression Baseline | 2 | 5 | 0 | 0
  Severe Major Depression Baseline | 0 | 0 | 0 | 0
  Major Depression Week 12 | 1 | 3 | 1 | 1
  Severe Major Depression Week 12 | 0 | 0 | 0 | 0
  Major Depression Week 24 | 2 | 0 | 0 | 0
  Severe Major Depression Week 24 | 0 | 0 | 0 | 0

9. Secondary Outcome: Participant Reported Quality of Life Assessment Using EQ-5D-5L Standardized Instrument
Description: The EQ-5D-5L is a self-administered general measure of health outcome applicable to a wide range of health conditions and treatments.The EQ-5D-5L measures quality of life in 5 dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. Each is rated in 5 levels from no problems/pain/anxiety to being unable/extreme pain/extreme anxiety. The responses for each category are summarized by treatment and visit with frequencies and percentages reporting each level.
Time Frame: Baseline and weeks 12, 24
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Participants
  No problem Walking Baseline | 1 | 0 | 1 | 2
  Slight Problem Walking Baseline | 1 | 2 | 2 | 1
  Moderate Problem Walking Baseline | 8 | 7 | 0 | 1
  Severe Problem Walking Baseline | 3 | 2 | 0 | 0
  Unable to Walk Baseline | 0 | 1 | 0 | 0
  No problem washing or dressing Baseline | 1 | 3 | 3 | 3
  Slight problem washing or dressing baseline | 1 | 3 | 0 | 1
  Moderate problem washing or dressing baseline | 10 | 5 | 0 | 0
  Severe problem washing or dressing baseline | 1 | 1 | 0 | 0
  Unable to wash or dress baseline | 0 | 0 | 0 | 0
  No problem doing usual activities Baseline | 0 | 0 | 0 | 1
  Slight problem doing usual activities Baseline | 0 | 1 | 2 | 2
  Moderate problem doing usual activities baseline | 10 | 5 | 1 | 1
  Severe problem doing usual activities baseline | 3 | 6 | 0 | 0
  Unable to do usual activities baseline | 0 | 0 | 0 | 0
  No pain or discomfort baseline | 0 | 0 | 0 | 0
  Slight pain or discomfort baseline | 0 | 0 | 1 | 2
  Moderate pain or discomfort baseline | 6 | 6 | 2 | 2
  Severe pain or discomfort baseline | 7 | 6 | 0 | 0
  Extreme pain or discomfort baseline | 0 | 0 | 0 | 0
  Not anxious or depressed baseline | 4 | 3 | 1 | 2
  Slightly anxious or depressed baseline | 5 | 4 | 2 | 2
  Moderately anxious or depressed baseline | 4 | 5 | 0 | 0
  Severely anxious or depressed baseline | 0 | 0 | 0 | 0
  Extremely anxious or depressed baseline | 0 | 0 | 0 | 0
  No problem Walking Week 12 | 1 | 0 | 1 | 1
  Slight Problem Walking Week 12 | 2 | 3 | 0 | 2
  Moderate Problem Walking Week 12 | 8 | 7 | 2 | 1
  Severe Problem Walking Week 12 | 2 | 2 | 0 | 0
  Unable to Walk Week 12 | 0 | 0 | 0 | 0
  No problem washing or dressing Week 12 | 2 | 3 | 1 | 3
  Slight problem washing or dressing Week 12 | 4 | 6 | 0 | 0
  Moderate problem washing or dressing week 12 | 5 | 3 | 2 | 1
  Severe problem washing or dressing Week 12 | 2 | 0 | 0 | 0
  Unable to wash or dress Week 12 | 0 | 0 | 0 | 0
  No problem doing usual activities Week 12 | 1 | 0 | 0 | 1
  Slight problem doing usual activities Week 12 | 4 | 3 | 1 | 1
  Moderate problem doing usual activities Week 12 | 4 | 6 | 1 | 2
  Severe problem doing usual activities Week 12 | 4 | 3 | 1 | 0
  Unable to do usual activities Week 12 | 0 | 0 | 0 | 0
  No pain or discomfort Week 12 | 0 | 0 | 0 | 0
  Slight pain or discomfort Week 12 | 0 | 1 | 0 | 1
  Moderate pain or discomfort Week 12 | 11 | 9 | 2 | 2
  Severe pain or discomfort Week 12 | 2 | 1 | 1 | 1
  Extreme pain or discomfort Week 12 | 0 | 1 | 0 | 0
  Not anxious or depressed Week 12 | 7 | 7 | 1 | 3
  Slightly anxious or depressed Week 12 | 2 | 4 | 0 | 0
  Moderately anxious or depressed Week 12 | 4 | 1 | 2 | 1
  Severely anxious or depressed Week 12 | 0 | 0 | 0 | 0
  Extremely anxious or depressed Week 12 | 0 | 0 | 0 | 0
  No problem Walking Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  No problem Walking Week 24 | 2 | 1 | 0 | 1
  Slight Problem Walking Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Slight Problem Walking Week 24 | 2 | 4 | 1 | 2
  Moderate Problem Walking Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Moderate Problem Walking Week 24 | 5 | 1 | 1 | 0
  Severe Problem Walking Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Severe Problem Walking Week 24 | 1 | 1 | 0 | 0
  Unable to Walk Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Unable to Walk Week 24 | 0 | 1 | 0 | 0
  No problem washing or dressing Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  No problem washing or dressing Week 24 | 3 | 2 | 1 | 2
  Slight problem washing or dressing Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Slight problem washing or dressing Week 24 | 3 | 4 | 0 | 1
  Moderate problem washing or dressing Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Moderate problem washing or dressing Week 24 | 3 | 0 | 1 | 0
  Severe problem washing or dressing Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Severe problem washing or dressing Week 24 | 1 | 2 | 0 | 0
  Unable to washing or dressing Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Unable to washing or dressing Week 24 | 0 | 0 | 0 | 0
  No problem doing usual activities Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  No problem doing usual activities Week 24 | 1 | 0 | 1 | 1
  Slight problem doing usual activities Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Slight problem doing usual activities Week 24 | 2 | 5 | 0 | 1
  Moderate problem doing usual activities Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Moderate problem doing usual activities Week 24 | 4 | 1 | 1 | 1
  Severe problem doing usual activities Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Severe problem doing usual activities Week 24 | 2 | 2 | 0 | 0
  Unable to do usual activities Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Unable to do usual activities Week 24 | 1 | 0 | 0 | 0
  No pain or discomfort Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  No pain or discomfort Week 24 | 0 | 0 | 0 | 1
  Slight pain or discomfort Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Slight pain or discomfort Week 24 | 1 | 4 | 1 | 1
  Moderate pain or discomfort Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Moderate pain or discomfort Week 24 | 5 | 1 | 1 | 1
  Severe pain or discomfort Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Severe pain or discomfort Week 24 | 4 | 3 | 0 | 0
  Extreme pain or discomfort Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Extreme pain or discomfort Week 24 | 0 | 0 | 0 | 0
  Not anxious or depressed Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Not anxious or depressed Week 24 | 4 | 5 | 1 | 2
  Slightly anxious or depressed Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Slightly anxious or depressed Week 24 | 3 | 0 | 1 | 1
  Moderately anxious or depressed Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Moderately anxious or depressed Week 24 | 3 | 3 | 0 | 0
  Severely anxious or depressed Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Severely anxious or depressed Week 24 | 0 | 0 | 0 | 0
  Extremely anxious or depressed Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Extremely anxious or depressed Week 24 | 0 | 0 | 0 | 0

10. Secondary Outcome: Participant Reported Quality of Life Assessment Using Visual Analog Scale (EQ-5D-5L Standardized Instrument)
Description: The EQ-5D-5L is a self-administered general measure of health outcome applicable to a wide range of health conditions and treatments. The visual analog scale (VAS) rates the subject's health on a 0-100 scale from the worst imaginable health state to the best imaginable health state.
Time Frame: Baseline to 12 and 24 week visit
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale
  Week 12 visit | 5.5 (11.45) | 3.2 (25.89) | -17.7 (12.01) | -6.3 (7.97)
  Week 24 visit | 4.5 (18.68) | 8.4 (28.57) | -4.5 (13.44) | 0.3 (5.86)

11. Secondary Outcome: Digit Symbol Substitution Test
Description: Overall neuropsychological function is assessed using the DSST, a test that is sensitive to brain damage, dementia, age, and depression, and is a widely used instrument for measuring the neuropsychological effects of opioid therapy. The digits (1-9) are paired with symbols, and the test consists of matching the symbol for a series of digits as fast as possible. Score is number of correct symbols in 90 seconds. A decrease from baseline detects deterioration in processing speed. An increase from baseline detects improvement in processing speed.
Time Frame: Change from Baseline to 12 and 24 week visit
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a test
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a test
  Week 12 from baseline | 7.8 (8.23) | 6.1 (10.22) | 3.3 (7.64) | 0.00 (4.83)
  Week 24 from baseline | 8.9 (8.41) | 0.1 (12.84) | -6.0 (5.66) | -3.3 (7.64)

12. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The Patient Global Impression of Change (PGIC) is a self-administered questionnaire that assesses the participant's level of improvement/worsening from the beginning to the end of treatment. Participants are asked to select the category of change that most closely describes any change experienced in the pain of their painful areas from the beginning of the Blinded Structured Opioid Discontinuation Period to Week 12 and to Week 24. The scale has levels describing change as: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Time Frame: Baseline to 12 and 24 week visit
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Participants
  Very much improved Week 12 | 0 | 0 | 0 | 0
  Much improved Week 12 | 3 | 1 | 0 | 1
  Minimally improved Week 12 | 8 | 5 | 1 | 1
  No change Week 12 | 1 | 3 | 0 | 0
  Minimally Worse Week 12 | 1 | 1 | 1 | 1
  Much Worse Week 12 | 0 | 2 | 0 | 1
  Very Much Worse Week 12 | 0 | 0 | 1 | 0
  Very much improved Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Very much improved Week 24 | 0 | 0 | 0 | 0
  Much improved Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Much improved Week 24 | 3 | 1 | 0 | 2
  Minimally improved Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Minimally improved Week 24 | 3 | 4 | 2 | 0
  No change Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  No change Week 24 | 3 | 1 | 0 | 0
  Minimally Worse Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Minimally Worse Week 24 | 1 | 2 | 0 | 0
  Much Worse Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Much Worse Week 24 | 0 | 0 | 0 | 1
  Very Much Worse Week 24: number analyzed (Participants) | 10 | 8 | 2 | 3
  Very Much Worse Week 24 | 0 | 0 | 0 | 0

13. Secondary Outcome: Sexual Function Measured Using the International Index of Erectile Function (IIEF) for Men and the Female Sexual Function Index (FSFI) for Women
Description: For the International Index of Erectile Function (IIEF)(15-items) each question is scored on a scale of 0 or 1 to 5, with 0 as no sexual attempts, 1 as the highest frequency, and 5 as the lowest, except where 1=1-2, 2=3-4, 3=5-6, 4=7-10 attempts, and 5=11 or more attempts. Missing responses are scored as 0. For the Female Sexual Function Index (FSFI)(19 items) each question is scored on a scale of 0-5 or 1-5. The FSFI examines the following 6 domains with minimum and maximum scores as indicated: desire(1.2-6.0), arousal(0-6.0), lubrication(0-6.0), orgasm(0-6.0), satisfaction(0.8-6.0), and pain(0-6.0). A computational formula sums the scores within each domain and multiplies that sum by a prescribed weighting factor: desire 0.6, arousal 0.3, lubrication 0.3, orgasm 0.4, satisfaction 0.4, pain 0.4. Higher scores indicate greater functionality. The single final score range is 2.0 to 36, which is reported as an average for each group of female study participants as change from baseline.
Time Frame: Change from Baseline to 12 and 24 week visit
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
Number analyzed (Participants) | 13 | 12 | 3 | 4
Score on a scale
  Male Erectile Function Week 12: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Erectile Function Week 12 | 2.0 (7.14) | -4.6 (10.26) | 4.0 (2.83) | 2.00 (7.07)
  Male Erectile Function Week 24: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Erectile Function Week 24 | 1.4 (13.56) | -0.4 (11.26) | 7.0 (9.90) | 4.5 (0.71)
  Male Orgasmic Function Week 12: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Orgasmic Function Week 12 | -1.0 (5.20) | -1.0 (4.24) | 0.5 (0.71) | 1.5 (0.71)
  Male Orgasmic Function Week 24: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Orgasmic Function Week 24 | -0.6 (7.33) | 0.4 (4.83) | 1.5 (0.71) | 2.0 (0.00)
  Male Sexual Desire Week 12: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Sexual Desire Week 12 | 2.2 (1.30) | 1.0 (2.35) | 0.0 (0.00) | 0.0 (0.00)
  Male Sexual Desire Week 24: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Sexual Desire Week 24 | 1.8 (2.59) | 0.8 (1.64) | -1.5 (3.54) | 0.0 (1.41)
  Male Intercourse Satisfaction Week 12: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Intercourse Satisfaction Week 12 | -1.0 (5.20) | -1.4 (5.22) | 0.5 (0.71) | 0.0 (0.00)
  Male Intercourse Satisfaction Week 24: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Intercourse Satisfaction Week 24 | -1.0 (7.68) | 0.4 (5.41) | 2.0 (2.83) | 1.5 (0.71)
  Male Overall Satisfaction Week 12: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Overall Satisfaction Week 12 | 1.8 (1.79) | 1.4 (3.36) | 1.5 (2.12) | 0.5 (2.12)
  Male Overall Satisfaction Week 24: number analyzed (Participants) | 5 | 5 | 2 | 2
  Male Overall Satisfaction Week 24 | 3.4 (1.67) | 2.2 (2.05) | 0.0 (2.83) | 0.0 (1.41)
  Female Desire Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Desire Week 12 | 0.23 (1.280) | -0.86 (1.544) | 0.00 (0) | 0.30 (0.424)
  Female Desire Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Desire Week 24 | 0.48 (1.301) | -1.40 (1.510) |  | 0.00 (0)
  Female Arousal Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Arousal Week 12 | 0.38 (2.711) | -0.47 (1.614) | -6.00 (0) | 1.35 (0.636)
  Female Arousal Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Arousal Week 24 | 1.80 (0.561) | -0.90 (1.559) |  | 0.90 (0)
  Female Lubrication Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Lubrication Week 12 | 0.00 (2.368) | 0.94 (1.514) | -3.60 (0) | 0.30 (0.000)
  Female Lubrication Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Lubrication Week 24 | 0.30 (2.205) | 0.30 (0.520) |  | 0 (0)
  Female Orgasm Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Orgasm Week 12 | -0.05 (2.216) | 0.91 (2.650) | -4.40 (0) | 0.20 (0.283)
  Female Orgasm Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Orgasm Week 24 | 0.40 (3.007) | 0.27 (0.462) |  | -0.40 (0)
  Female Satisfaction Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Satisfaction Week 12 | -0.10 (0.849) | -0.40 (3.046) | -0.40 (0) | 0.0 (0.00)
  Female Satisfaction Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Satisfaction Week 24 | -0.72 (1.277) | -0.67 (1.155) |  | 0.00 (0)
  Female Pain Week 12: number analyzed (Participants) | 8 | 7 | 1 | 2
  Female Pain Week 12 | 0.65 (3.312) | 2.69 (2.589) | -3.20 (0) | -0.40 (1.131)
  Female Pain Week 24: number analyzed (Participants) | 5 | 3 | 0 | 1
  Female Pain Week 24 | 0.88 (3.411) | 0.80 (1.386) |  | 0.40 (0)

ADVERSE EVENTS:
Time Frame: Up to 34 Weeks Post Randomization
Groups:
- Structured Discontinuation Opioid Therapy Optimal Responder: Structured discontinuation of opioid therapy (morphine sulfate ER, oxycodone ER, oxymorphone ER), Optimal Respond
Arm/Group | Structured Discontinuation Opioid Therapy Suboptimal Responder | Continuation of Opioid Therapy Suboptimal Responder | Structured Discontinuation Opioid Therapy Optimal Responder | Continuation of Opioid Therapy Optimal Responder
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/12 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 9/13 | 7/12 | 2/3 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Structured Discontinuation Opioid Therapy Suboptimal Responder (N=13) | Continuation of Opioid Therapy Suboptimal Responder (N=12) | Structured Discontinuation Opioid Therapy Optimal Responder (N=3) | Continuation of Opioid Therapy Optimal Responder (N=4)
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Structured Discontinuation Opioid Therapy Suboptimal Responder (N=13) | Continuation of Opioid Therapy Suboptimal Responder (N=12) | Structured Discontinuation Opioid Therapy Optimal Responder (N=3) | Continuation of Opioid Therapy Optimal Responder (N=4)
Drug Screen Positive (Investigations) | 2 | 1 | 0 | 0
Urine Alcohol Test Positive (Investigations) | 1 | 1 | 0 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perineal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Haematotympanum (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Ear Pain (General disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated because it could not recruit the planned study population. Randomized study participants were too few to show changes in pain intensity scores or clinical effects. The safety profile reflects current prescribing information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT02741076/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02741076/SAP_001.pdf